CLINICAL TRIAL: NCT01260870
Title: European Study of POBA Versus Cotavance Paclitaxel Coated Balloon for the Treatment of Infrapopliteal Lesions in Critical Limb Ischemia
Brief Title: European Study of POBA Versus Cotavance(R) Paclitaxel Coated Balloon for the Treatment of Infrapopliteal Lesions in Critical Limb Ischemia (EURO CANAL)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Bayer terminated the program and sold the IP to Medronic
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EURO CANAL
Record Dates: First submitted 2010-12-13; First posted 2010-12-15 (Estimated); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: PAD; Infrapopliteal Lesions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cotavance (Experimental)
  Interventions: Device: Cotavance Paclitaxel Coated Balloon
- Standard balloon angioplasty (Active Comparator): POBA
  Interventions: Device: Standard balloon angioplasty

INTERVENTIONS:
Device: Cotavance Paclitaxel Coated Balloon
  Other Names: DEB
  Arms: Cotavance
Device: Standard balloon angioplasty
  Other Names: POBA
  Arms: Standard balloon angioplasty

SUMMARY:
To evaluate the procedural safety and to identify and characterize therapeutic and functional endpoint assessments in subjects with documented critical limb ischemia who received treatment with the Cotavance Paclitaxel-Coated Balloon vs. those who received POBA only.

ELIGIBILITY:
Inclusion Criteria:

- Subjects with CLI

Exclusion Criteria:

* Participation in another research trial
* Medical conditions the study doctor will assess

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-08-15 (Actual); Primary Completion 2013-07-15 (Actual); Study Completion 2013-07-15 (Actual)

PRIMARY OUTCOMES:
Evaluate procedural safety | 30 days

SECONDARY OUTCOMES:
Identify and characterize therapeutic and functional endpoint assessments | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (6):
- Medical University, Graz, Austria
- Belgium (2):
  - AZ St.-Blasius Hospital, Dendermonde
  - University Hospital, Ghent
- Switzerland (2):
  - University Hospital, Bern
  - University Hospital, Zurich
- St. George's Hospital, London, United Kingdom